CLINICAL TRIAL: NCT00956748
Title: N-Acetylcysteine as an Adjunct for Refractory Chronic Suppurative Otitis Media
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of staff, time, and resources
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Dr Brian Westerberg, Clinical Professor, Department of Surgery, UBC Otology & Neurotology, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H09-00953
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Otitis Media; Otorrhea
Keywords: chronic suppurative otitis media with persistent otorrhea
MeSH Terms: conditions — Otitis Media | interventions — Ciprofloxacin; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprodex otic solution (Active Comparator): ciprofloxacin 0.3% / dexamethasone 0.1% otic solution
  Interventions: Drug: Ciprodex
- Ciprodex with 2% NAC (Experimental): Ciprodex otic solution (ciprofloxacin 0.3% / dexamethasone 0.1%) augmented with 2% N-acetylcysteine
  Interventions: Drug: Ciprodex and 2% NAC

INTERVENTIONS:
Drug: Ciprodex — Administer 3 to 5 drops tid for 14 days. Continue treatment for another 14 days if otorrhea persists.
  Other Names: ciprofloxacin 0.3% / dexamethasone 0.1%
  Arms: Ciprodex otic solution
Drug: Ciprodex and 2% NAC — Administer 3 to 5 drops tid for 14 days. Continue treatment for another 14 days if otorrhea persists.
  Other Names: Ciprodex with 2% N-Acetylcysteine
  Arms: Ciprodex with 2% NAC

SUMMARY:
Chronic suppurative otitis media (CSOM) can be particularly difficult to treat as a number of patients do not respond to routine antibiotic or surgical treatments. The current treatment involves administering combination antibiotic anti-inflammatory ear drops such as Ciprodex (ciprofloxacin 0.3% / dexamethasone 0.1%). Although most patients experience a relief of symptoms, a fraction of patients remain refractory to treatment. Recent findings suggest that the addition of N-acetylcysteine (0.5-2%) to Ciprodex is a superior treatment for otitis media with effusion compared to the use of Ciprodex alone.

DETAILED DESCRIPTION:
Chronic suppurative otitis media (CSOM) is the presence of symptoms, signs, and physical findings that can result in long-term damage to the middle ear as a result of infection or inflammation. The condition is defined as chronic drainage from the ear, lasting longer than 12 weeks, through a perforated tympanic membrane. Although the pathogenesis may result from the actions of inflammatory mediators and cytokines released following an infection, recent evidence also suggests that biofilm formation may be responsible for sustaining the inflammatory response that promotes the persistent effusion (1). These patients present a challenge to otolaryngologists because a number do not respond to typical oral and topical antibiotics.

N-acetylcysteine (NAC) is an antioxidant commonly used in the treatment of acetaminophen overdose, and has well documented mucolytic properties. In vitro, NAC has been shown to significantly inhibit the formation of bacterial biofilms when used alone or enhance the antimicrobial effects of other drugs such as ciprofloxacin (3), fosfomycin and tigecycline when used in combination (4-6). The application of NAC to the middle ear in patients with tympanostomy tubes has been shown to increase tube longevity, and decrease the replacement of tubes, recurrence of infection, tympanosclerosis, and subsequent physician visits (7). Recent findings from a case series suggest that the addition of N-acetylcysteine (NAC) to Ciprodex otic solution is a superior treatment for chronic otitis media compared to Ciprodex alone (3). Although the practice of supplementing Ciprodex otic solution, a standard pharmacologic treatment for otitis media, with NAC in order to treat patients with difficult infections holds therapeutic promise, the efficacy of the treatment has not been objectively assessed in a controlled study to date in a patient population of adequate size.

The purpose of this study will be to assess the efficacy of Ciprodex augmented with NAC compared to Ciprodex alone in a blinded study in subjects for whom other therapies for a chronically draining ear have been ineffective.

Hypothesis:

The cessation of otorrhea is expected to be achieved in a greater number of subjects with otorrhea treated with Ciprodex otic solution supplemented with NAC compared to Ciprodex alone. We expect that patients treated with Ciprodex augmented with NAC will experience an earlier cessation of symptoms and a longer duration of complete response following treatment.

Justification:

The current pharmacologic treatment for CSOM involves combination antibiotic anti-inflammatory otic drops. Ciprodex (ciprofloxacin 0.3% / dexamethasone 0.1%) has been shown to be safe and effective in both children and adults with ear infections. Although most patients experience a relief of symptoms, clinical data from various studies show 10-15% patients do not respond to treatment (2). Recent findings suggest that the addition of N-acetylcysteine (NAC) to Ciprodex otic solution is a superior treatment for chronic otitis media compared to Ciprodex alone (3).

Objectives:

The specific aim of this project is to compare the effect of Ciprodex otic solution alone with the use of Ciprodex augmented with 1.25% NAC in a randomized double-blind trial.

Research Method:

Patients who have experienced at least 1 month of continuous daily otorrhea despite treatment will be recruited from tertiary otology/neurotology clinics. Patient information, including previous failed interventions, duration of otorrhea, baseline audiometry, and existing medical conditions will be documented prior to initiating treatment.

Subjects will be randomly assigned to one of the two treatment groups and instructed to administer 3 drops three times daily in the affected ear for 14 days. One group will use standard Ciprodex solution; the second group will use Ciprodex to which 0.5mL of 20% NAC was added to the 7.5mL bottle (final concentration 1.25%)

Follow-up visits will be scheduled in 2 week intervals, where patients will undergo audiometry re-assessment and treatment progress will be monitored by history and binocular microscopy. Compliance to treatment will be confirmed during follow-up visits and patients will be provided fresh otic solution for a further 14 days if the discharge persists, to a maximum duration of therapy of 8 weeks. During this period patients will be assessed every 2 weeks, as is currently the standard treatment. Potential adverse reactions such as otalgia, tinnitus, ear fullness, or vertigo will also be documented at each visit. After a maximum of 8 weeks of treatment, patients who continue to experience otorrhea will undergo alternative treatment regimens which may include oral or topical antibiotics, or surgery. Patients who have been successfully treated will be monitored at 4 to 6 months to assess whether a complete and durable cessation of otorrhea has been achieved.

Randomization of the drugs will be performed by the hospital site pharmacists prior to dispensing the solution to subjects. Random number lists will be generated and randomization performed in blocks of 4 through the St. Paul's Hospital Pharmacy. The Principle Investigator will have access to the database should an emergency situation arise.

Statistical Analysis:

Statistical analysis including two-tailed paired Student's t tests will be performed to compare the treatment duration required before patients experience a cessation of otorrhea for each of the two treatment groups. Thirty patients (15 per treatment group) are expected to be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* continuous otorrhea for a duration of greater than 6 months
* at least 2 previous treatment regimes for otitis media, which may include topical or oral antibiotics, myringotomy or tympanostomy, and surgery

Exclusion Criteria:

* existing cholesteatoma
* known allergy to ciprofloxacin, dexamethasone, or N-acetylcysteine
* patients who are unlikely to adhere to the treatment regime and follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
cessation of otorrhea | 4 weeks

SECONDARY OUTCOMES:
durable cessation of otorrhea | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Westerberg, MD, Principal Investigator — St. Paul's Hospital Rotary Hearing Clinic
Locations (1):
- St. Paul's Hospital BC Rotary Hearing & Balance Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fergie N, Bayston R, Pearson JP, Birchall JP. Is otitis media with effusion a biofilm infection? Clin Otolaryngol Allied Sci. 2004 Feb;29(1):38-46. doi: 10.1111/j.1365-2273.2004.00767.x. PMID 14961850
- [Background] Wall GM, Stroman DW, Roland PS, Dohar J. Ciprofloxacin 0.3%/dexamethasone 0.1% sterile otic suspension for the topical treatment of ear infections: a review of the literature. Pediatr Infect Dis J. 2009 Feb;28(2):141-4. doi: 10.1097/INF.0b013e31818b0c9c. PMID 19116600
- [Background] Choe WT, Murray MT, Stidham KR, Roberson JB. N-Acetylcysteine as an adjunct for refractory ear infections. Otol Neurotol. 2007 Dec;28(8):1022-5. doi: 10.1097/MAO.0b013e318155a4d3. PMID 17898673
- [Background] Perez-Giraldo C, Rodriguez-Benito A, Moran FJ, Hurtado C, Blanco MT, Gomez-Garcia AC. Influence of N-acetylcysteine on the formation of biofilm by Staphylococcus epidermidis. J Antimicrob Chemother. 1997 May;39(5):643-6. doi: 10.1093/jac/39.5.643. PMID 9184365
- [Background] Marchese A, Bozzolasco M, Gualco L, Debbia EA, Schito GC, Schito AM. Effect of fosfomycin alone and in combination with N-acetylcysteine on E. coli biofilms. Int J Antimicrob Agents. 2003 Oct;22 Suppl 2:95-100. doi: 10.1016/s0924-8579(03)00232-2. PMID 14527779
- [Background] Aslam S, Trautner BW, Ramanathan V, Darouiche RO. Combination of tigecycline and N-acetylcysteine reduces biofilm-embedded bacteria on vascular catheters. Antimicrob Agents Chemother. 2007 Apr;51(4):1556-8. doi: 10.1128/AAC.00893-06. Epub 2007 Jan 12. PMID 17220399
- [Background] Ovesen T, Felding JU, Tommerup B, Schousboe LP, Petersen CG. Effect of N-acetylcysteine on the incidence of recurrence of otitis media with effusion and re-insertion of ventilation tubes. Acta Otolaryngol Suppl. 2000;543:79-81. doi: 10.1080/000164800454044. PMID 10908985